CLINICAL TRIAL: NCT04532853
Title: Optimizing Maintenance Therapy in COPD Patients: Real-world Observational Study of Peak Inspiratory Flow Rate, Inhalation Technique, and Medication Adherence
Brief Title: Optimizing Maintenance Therapy in COPD Patients
Acronym: PIFOTAL
Status: Completed | Type: Observational
Sponsor: General Practitioners Research Institute (Network)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: GPRI20103
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: COPD
Keywords: COPD Exacerbations; Primary Care; Inhalation medication; Epidemiology; Treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients

SUMMARY:
Background: Effectiveness of maintenance therapy for COPD with Dry Powder Inhalers (DPIs) requires an optimal Peak Inspiratory Flow Rate (PIFR), a proper inhalation technique and adequate medication adherence from patients. Recent studies have suggested that patients with reduced peak inspiratory flow may have worse COPD-related symptom burden and increased risk of COPD-related hospitalizations. However, in primary care, little is known about how many COPD patients have suboptimal PIFR. Furthermore, there is a paucity of knowledge concerning the associations of PIFR, inhalation technique and medication adherence with the effectiveness of maintenance therapy.

Objective: To examine associations of PIFR, inhalation technique, and medication adherence with health status and disease, exacerbations, and healthcare resource utilization in patients with COPD receiving maintenance treatment with dry powder inhalers.

Study design: Cross-sectional observational study in five European countries*.

Study population: COPD patients aged 40 years or older who have received COPD maintenance therapy through DPIs in the past 3 months or longer.

Main study parameters: Health status as measured with the Clinical COPD Questionnaire (CCQ), COPD Assessment Test (CAT), number of exacerbations, an assessment of PIFR, inhalation technique errors, medication adherence, healthcare resource utilization (HCRU), medication use and demographic and clinical covariates.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: No significant burden from participating is expected. Risk of participating is deemed negligible. In addition, patients may benefit from participating. Specifically, patients who manifest inhalation errors, will receive a tailored inhalation instruction to remediate their inhalation errors. The impact of this instruction will not be evaluated in any way, therefore it should not be seen as an intervention.

* If the preplanned number of patients cannot be included also because of national outbreaks of SARS-COV-2 resulting in travel restrictions, participation will be sought from researchers from three other European countries

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of COPD;
* Age ≥ 40;
* Use of maintenance therapy through a DPI in the last 3 months or longer
* Sufficient investigator-assessed decision-making capacity to provide informed consent (patients will not be invited if they have acute psychotic disorders, severe pervasive developmental disorders / severe intellectual disability or advanced neurodegenerative disease)

Exclusion Criteria:

* An exacerbation in the past 6 weeks (as this requires a patient to recover)
* Life threatening disease and life expectancy < 6 months (as inclusion of these patients is unethical)
* Participation in a randomized clinical trial on COPD medication

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients aged forty years and older and who are treated with DPIs as a maintenance therapy
Sampling Method: Non-Probability Sample
Enrollment: 1434 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Clinical COPD Questionnaire | past 7 days (counted from day of study visit)
  Self reported health status of COPD
COPD Assessment Test (CAT) | past 7 days (counted from day of study visit) [Note that the CAT has no explicit time frame]
  Self reported health status of COPD

SECONDARY OUTCOMES:
COPD Exacerbations | past 12 months (counted from day of study visit)
  Self reported
Healthcare resource utilization | past 6 months (counted from day of study visit)
  Of primary care (consultations with GPs and primary care nurse), of secondary care (consultations with registrars or medical specialists in outpatient clinics, emergency departments, rate and duration of hospitalizations, and chest imaging/x-rays), of other healthcare provision (lung function technicians, physiotherapists, dietitians, and psychologists), as well as laboratory assessments and medication use.

CONTACTS AND LOCATIONS:
Overall Officials: Janwillem Kocks, MD, PhD, Principal Investigator — General Practitioners Research Institute
Locations (6):
- Woolcock Institute of Medical Research, University of Sydney, Sydney, Australia
- University of Crete, Heraklion, Greece
- GPRI, Groningen, Netherlands
- Medical University of Silesia, Katowice, Poland
- Center Health Regional Administration (ARS Centro), Aveiro, Portugal
- Ibsalut, Soller, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kocks J, Bosnic-Anticevich S, van Cooten J, Correia de Sousa J, Cvetkovski B, Dekhuijzen R, Dijk L, Garcia Pardo M, Gardev A, Gawlik R, van der Ham I, Janse Y, Lavorini F, Maricoto T, Meijer J, Metz B, Price D, Roman Rodriguez M, Schuttel K, Stoker N, Tsiligianni I, Usmani O, Voorham J, Leving MT. Identifying critical inhalation technique errors in Dry Powder Inhaler use in patients with COPD based on the association with health status and exacerbations: findings from the multi-country cross-sectional observational PIFotal study. BMC Pulm Med. 2023 Aug 17;23(1):302. doi: 10.1186/s12890-023-02566-6. PMID 37592263
- [Derived] Leving MT, Bosnic-Anticevich S, van Cooten J, de Sousa JC, Cvetkovski B, Dekhuijzen R, Dijk L, Pardo MG, Gardev A, Gawlik R, van der Ham I, Janse Y, Lavorini F, Maricoto T, Meijer J, Metz B, Price D, Roman-Rodriguez M, Schuttel K, Stoker N, Tsiligianni I, Usmani O, Emerson-Stadler R, Kocks JWH. Clinical recommendations for dry powder inhaler use in the management of COPD in primary care. NPJ Prim Care Respir Med. 2022 Dec 27;32(1):59. doi: 10.1038/s41533-022-00318-3. PMID 36575175
- [Derived] Leving M, Wouters H, de la Hoz A, Bosnic-Anticevich S, Dekhuijzen R, Gardev A, Lavorini F, Meijer J, Price D, Rodriguez MR, Tsiligianni I, Usmani O, Wijnsma B, Kocks J. Impact of PIF, Inhalation Technique and Medication Adherence on Health Status and Exacerbations in COPD: Protocol of a Real-World Observational Study (PIFotal COPD Study). Pulm Ther. 2021 Dec;7(2):591-606. doi: 10.1007/s41030-021-00172-7. Epub 2021 Sep 17. PMID 34533772